CLINICAL TRIAL: NCT02421315
Title: Overlapping Neural Circuits Implicated in Pediatric OCD
Brief Title: Overlapping Neural Circuits in Pediatric OCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Rachel Marsh, Irving Philips Professor of Medical Psychology (in Child Psychology), New York State Psychiatric Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 7006; R21MH101441 (NIH)
Record Dates: First submitted 2015-04-09; First posted 2015-04-20 (Estimated); Results first posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Obsessive Compulsive Disorder
Keywords: OCD; Functional Magnetic Resonance Imaging (fMRI); Magnetic Resonance Imaging (MRI)
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Participants With Obsessive-compulsive Disorder (OCD) (Experimental): Children and adolescents who meet DSM-IV diagnostic criteria for OCD and had clinically significant obsessive-compulsive symptoms (CY-BOCS score>15). Comorbid anxiety disorders, but no other lifetime psychiatric diagnoses, were permitted in the OCD group as long as OCD was the primary diagnosis. Participants were unmedicated and had not received a full course of CBT with exposure and response prevention for OCD prior to their participation in the study. Following baseline assessment and scan, patients with OCD underwent a course of manualized treatment of CBT with E/RP adapted for pediatric OCD delivered by a licensed clinical psychologist or advanced supervised graduate student in clinical psychology at the NYSPI.
  Interventions: Behavioral: CBT treatment for OCD based on Exposure & Response Prevention (EX/RP) and when indicated medication treatment
- Healthy Control (HC) Participants (No Intervention): Healthy control (HC) participants matched on age and sex with the OCD group. HC participants had no lifetime psychiatric disorders. HC participants were assessed and scanned at baseline and again after 12-16 weeks.

INTERVENTIONS:
Behavioral: CBT treatment for OCD based on Exposure & Response Prevention (EX/RP) and when indicated medication treatment — CBT treatment consisted of 12-16 hour-long sessions. For exceptional cases not showing clinical improvement after six CBT treatment sessions, complementary pharmacological treatment (SSRI) was offered as part of our treatment protocol. CBT for OCD involves gradually exposing patients to anxiety provoking stimuli while having patients refrain from engaging in compulsive rituals and/or avoidance behaviors. There are three major components of CBT treatment for OCD, specifically: (1) exposure to anxiety provoking stimuli, (2) response prevention, and (3) cognitive techniques intended to decrease anxiety during the exposure and response prevention processes.
  Arms: Participants With Obsessive-compulsive Disorder (OCD)

SUMMARY:
The purpose of this study is to examine the brain functioning of children and adolescent with OCD before and after treatment with Exposure and Response Prevention (EXRP) therapy.

DETAILED DESCRIPTION:
The capacity to coordinate thoughts and actions to execute goal-directed behaviors (cognitive control) and the capacity to anticipate, respond to, and learn from reward (reward processing) are key processes for human behavior. Dysfunction in these processes has been hypothesized to contribute to repetitive thoughts and behaviors in many disorders, including obsessive-compulsive disorder (OCD), Tourette Syndrome (TS), and eating disorders. The investigators will use multimodal imaging to investigate neural circuits that support cognitive control and reward processing, using pediatric OCD as a model system. The short-term goal is to clarify how circuit-based abnormalities contribute to repetitive thoughts/behaviors; these data will inform future trans-diagnostic studies. The long-term goal is to identify control and reward circuit-abnormalities as targets for new trans-diagnostic treatments.

ELIGIBILITY:
Patient Inclusion Criteria:

* Participants must be 5-17 at the time of consent
* Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) Diagnosis of OCD as the principal problem
* Not on psychotropic medication and not receiving current psychotherapy for OCD
* Written informed assent by the participants (8 and older) and consent by the parent
* Participants and a parent/guardian must be able to read and understand English

Patient Exclusion Criteria:

* DSM-IV current diagnosis of major depressive disorder, attention-deficit hyperactivity disorder, Tourette's/Tic Disorder, or substance/alcohol abuse
* DSM-IV lifetime diagnosis of psychotic disorder, bipolar disorder, eating disorder, pervasive developmental disorder, or substance/alcohol abuse
* Active suicidal ideation
* Females who are pregnant or nursing
* Major medical or neurological problems
* Presence of metallic device or dental braces
* IQ<80
* A current or past diagnosis of pediatric autoimmune neuropsychiatric disorders associated with streptococcus (PANDAS)
* Individuals who are currently receiving CBT, other forms of psychotherapy, or psychotropic medications
* Individuals who have received a full course of CBT in the past
* A positive pregnancy test
* Positive urine screen for illicit drugs
* Inability of participant or parent/guardian to read or understand English

Healthy Control Inclusion Criteria:

* Participants must be 5-17 at the time of consent
* Written informed assent by the participants (8 and older) and consent by the parent
* Participants and a parent/guardian must be able to read and understand English

Healthy Control Exclusion Criteria:

* Any current or lifetime psychiatric diagnosis
* Active suicidal ideation
* Females who are pregnant or nursing
* Major medical or neurological problems
* Presence of metallic device or dental braces
* IQ<80
* A current or past diagnosis of pediatric autoimmune neuropsychiatric disorders associated with streptococcus (PANDAS)
* A positive pregnancy test
* Positive urine screen for illicit drugs
* Inability of participant or parent/guardian to read or understand English

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2014-10; Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Marsh, Ph.D., Principal Investigator — New York Psychiatric Institute
Locations (1):
- NY State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Wang Z, Fontaine M, Cyr M, Rynn MA, Simpson HB, Marsh R, Pagliaccio D. Subcortical shape in pediatric and adult obsessive-compulsive disorder. Depress Anxiety. 2022 Jun;39(6):504-514. doi: 10.1002/da.23261. Epub 2022 Apr 29. PMID 35485920
- [Derived] Lv D, Ou Y, Wang Y, Ma J, Zhan C, Yang R, Chen Y, Shang T, Jia C, Sun L, Zhang G, Sun Z, Li J, Wang X, Guo W, Li P. Altered Functional Connectivity Strength at Rest in Medication-Free Obsessive-Compulsive Disorder. Neural Plast. 2021 Sep 8;2021:3741104. doi: 10.1155/2021/3741104. eCollection 2021. PMID 34539777
- [Derived] Cyr M, Pagliaccio D, Yanes-Lukin P, Fontaine M, Rynn MA, Marsh R. Altered network connectivity predicts response to cognitive-behavioral therapy in pediatric obsessive-compulsive disorder. Neuropsychopharmacology. 2020 Jun;45(7):1232-1240. doi: 10.1038/s41386-020-0613-3. Epub 2020 Jan 17. PMID 31952071
- [Derived] Pagliaccio D, Cha J, He X, Cyr M, Yanes-Lukin P, Goldberg P, Fontaine M, Rynn MA, Marsh R. Structural neural markers of response to cognitive behavioral therapy in pediatric obsessive-compulsive disorder. J Child Psychol Psychiatry. 2020 Dec;61(12):1299-1308. doi: 10.1111/jcpp.13191. Epub 2019 Dec 31. PMID 31889307

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Obsessive-compulsive Disorder (OCD): Children and adolescents who meet DSM-IV diagnostic criteria for OCD and had clinically significant obsessive-compulsive symptoms (CY-BOCS score > 15). Comorbid anxiety disorders, but no other lifetime psychiatric diagnoses, were permitted in the OCD group as long as OCD was the primary diagnosis. Participants were unmedicated and had not received a full course of CBT with exposure and response prevention for OCD prior to their participation in the study. Following baseline assessment and scan, patients with OCD underwent a course of manualized treatment of CBT with E/RP adapted for pediatric OCD (March & Mulle, 1998) delivered by a licensed clinical psychologist or advanced supervised graduate student in clinical psychology at the NYSPI. CBT treatment consisted of 12-16 hour-long sessions. For exceptional cases not showing clinical improvement after six CBT treatment sessions, complementary pharmacological treatment (SSRI) was offered as part of our treatment protocol. CBT for OCD involves gradually exposing patients to anxiety provoking stimuli while having patients refrain from engaging in compulsive rituals and/or avoidance behaviors. There are three major components of CBT treatment for OCD, specifically: (1) exposure to anxiety provoking stimuli, (2) response prevention, and (3) cognitive techniques intended to decrease anxiety during the exposure and response prevention processes.
- Healthy Control (HC) Participants: Healthy control (HC) participants matched on age and sex with the OCD group. HC participants had no lifetime psychiatric disorders. HC participants were assessed and scanned at baseline .
Period: Overall Study
Arm/Group | Participants With Obsessive-compulsive Disorder (OCD) | Healthy Control (HC) Participants
Started | 28 | 27
Completed | 23 | 15
Not Completed | 5 | 12

BASELINE CHARACTERISTICS:
Groups:
- Healthy Control (HC) Participants: Healthy control (HC) participants matched on age and sex with the OCD group. HC participants had no lifetime psychiatric disorders. HC participants were assessed and scanned at baseline.
- Total: Total of all reporting groups
Arm/Group | Participants With Obsessive-compulsive Disorder (OCD) | Healthy Control (HC) Participants | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.14 (3.34) | 11.26 (3.23) | 11.69 (3.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 14 | 14 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 9 | 16
  Not Hispanic or Latino | 21 | 16 | 37
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 21 | 8 | 29
  More than one race | 4 | 9 | 13
  Unknown or Not Reported | 1 | 5 | 6
Region of Enrollment [Number; unit: participants]
  United States | 28 | 27 | 55
Full Scale Intelligence Quotient (FSIQ) [Mean (Standard Deviation); unit: T-Score] — The FSIQ is a score derived from administration of 4 selected subtests (vocabulary, similarities, block design, and matrix reasoning) from the Wechsler Abbreviated Intelligence Scale - Second Edition (WASI-II), to provide a measure of global level of general cognitive and intellectual functioning.
  Standard scores are normed with a population mean of 100 and standard deviation of 15.
  Interpretation of Standard Score Ranges in terms of Performance: >129=Superior;120-129=Very High; 110-119=Bright Normal Performance; 90-109=Average; 80-89=Low Average; 70-79=Borderline Mental Functioning.
  T-Score | 106.96 (16.20) | 109.59 (12.14) | 108.25 (13.95)

OUTCOME MEASURES:

1. Primary Outcome: Brain Activation Associated With the Resolution of Cognitive Conflict
Description: Task-based functional magnetic resonance imaging (fMRI) will be acquired from children and adolescents diagnosed with OCD and healthy comparison subjects (HCs) during their performance of a Simon Spatial Compatibility Task.
  In each trial, participants are presented with a leftward or rightward pointing arrow that is either congruent or incongruent with their position (left or right) on the screen. Participants are instructed to respond as quickly and accurately as possible to the direction in which the arrow was pointing by pressing a button on a response box using the index finger for left and the middle finger for right. Brain activation during the resolution of cognitive conflict is computed by contrasting blood-oxygen-level-dependent (BOLD) signal during Incongruent versus Congruent trials. BOLD signal is expressed in arbitrary units (A.U.s).
Time Frame: single time point: baseline
Population: Only participants with usable fMRI data were included in these analyses. One participant with OCD and 4 HC participants were excluded because of missing fMRI data.
Measure: Mean (Standard Deviation); unit: Arbitrary units
Arm/Group | Participants With Obsessive-compulsive Disorder (OCD) | Healthy Control (HC) Participants
Number analyzed (Participants) | 27 | 23
Arbitrary units | .7 (.2) | .59 (.2)
Statistical Analysis 1: Comparison: Participants With Obsessive-compulsive Disorder (OCD) vs Healthy Control (HC) Participants; We hypothesized that compared to HC, children and adolescents with OCD would have increased activation in subcortical structures (insula, and putamen) comprising a right hemisphere dorsal frontostriatal circuit; Test type: Other — a t-test comparing groups in a specific region-of-interest (ROI); the insula; p = 0.0585, t-test, 2 sided; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.004 to 0.224], Standard Error of Mean 0.057

2. Secondary Outcome: Functional Connectivity
Description: Functional magnetic resonance imaging (fMRI) will be acquired from children and adolescents diagnosed with OCD and healthy comparison subjects (HCs) at baseline and after approximately 16-20 weeks (i.e., post-treatment for the participants with OCD). The whole brain is divided in 352 brain regions comprised of 333 cortical surface (Gordon et al. Cereb Cortex 2016;26:288-303) and 19 subcortical (Fischl et al. Neuron 2002;53:341-55) parcellated regions. FC-strength (average of Fisher-r-to-Z transformed Pearson correlation coefficients) between each region was computed.
  Values >0 indicate regions are positively connected (synchronized), with larger values indicating stronger connection. Values <0 indicate regions are negatively connected (inversely synchronized), with more negative values stronger negative connection. A value of 0 indicates that the regions are not connected.
Time Frame: single time point: Baseline
Population: Only participants with usable fMRI data were included in these analyses. Three participants with OCD and 4 HC participants were excluded because of missing fMRI data.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Participants With Obsessive-compulsive Disorder (OCD) | Healthy Control (HC) Participants
Number analyzed (Participants) | 25 | 23
arbitrary units | -0.312768356 (0.223710827) | 0.182360856 (0.230155947)
Statistical Analysis 1: Comparison: Participants With Obsessive-compulsive Disorder (OCD) vs Healthy Control (HC) Participants; Whole-Brain Connectome-Level Analyses were performed on the FC-strength indices between 352 regions. Edge-wise functional connectivity analyses was then be conducted across the resulting matrix comprised of 352 nodes and 123,904 edges, using the Network-Based Statistics (NBS) Toolbox. We hypothesized that youth with OCD would show altered FC between task-control circuit regions; Test type: Superiority — We selected 'arbitrary units' as the unit of measure here because we are looking at connectivity strengths; p = .037, t-test, 1 sided — NBS controls for family-wise error rate using permutation testing to identify components or "clusters" of contiguous region-to-region connections. A statistical threshold of p<.05 with 20,000 permutations was used; Mean Difference (Final Values) = 0.49512921, Standard Error of Mean 0.06553315 — Direction of the comparison: HC>OCD
Statistical Analysis 2: Comparison: Participants With Obsessive-compulsive Disorder (OCD); Separate cross-lagged panel models were computed in the OCD group for the three functional connections that differed significantly across groups at baseline (see Statistical Analysis 1). These models were constructed using IBM SPSS Amos (v.23) to test for directional relationships between OCD symptoms and FC pre- to post-treatment in the OCD patients. CY-BOCS total scores at each time point were used as the OCD symptoms measure; Test type: Other; p < .05, Regression, Linear; Slope = -.521

3. Secondary Outcome: Brain Gray Matter Thickness
Description: Structural MRI will be acquired from children and adolescents diagnosed with OCD and healthy comparison subjects (HCs). Regional cortical thickness will be computed in the inferior frontal gyrus
Time Frame: Single time point: Baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Participants With Obsessive-compulsive Disorder (OCD) | Healthy Control (HC) Participants
Number analyzed (Participants) | 28 | 27
mm | 3 (0.2) | 2.89 (0.2)
Statistical Analysis 1: Comparison: Participants With Obsessive-compulsive Disorder (OCD) vs Healthy Control (HC) Participants; Test type: Superiority; p = 0.0464, t-test, 2 sided; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [0.0018 to 0.218]

4. Secondary Outcome: Structural Connectivity (Streamline Counts)
Description: Magnetic Resonance Imaging (MRI) with Diffusion Tensor Imaging (DTI) will be acquired from children and adolescents diagnosed with OCD and healthy comparison subjects (HCs). A structural connectivity matrix is estimated for each participant using the standard MRtrix3 preprocessing pipeline, yielding 164x164 symmetrical streamline count matrix for each participant using the FreeSurfer segmentations/parcellations noted above (148 cortical, 14 subcortical regions, and the left and right cerebellum). Using this approach, streamline count between brain regions is proportional to the cross-sectional area of white matter fibers connecting those regions. Thus, streamline count is a biologically plausible metric of "structural connectivity" proposed to represent the communication 'bandwidth' between regions.
Time Frame: Single time point (baseline)
Population: Only participants with usable DTI data were included in these analyses. Three participants with OCD and 2 HC participants were excluded because of missing DTI data.
Measure: Mean (Standard Deviation); unit: streamlines
Units Other Than Participants: streamlines
Arm/Group | Participants With Obsessive-compulsive Disorder (OCD) | Healthy Control (HC) Participants
Number analyzed (Participants) | 25 | 25
Number analyzed (streamlines) | 26896 | 26896
streamlines | 227.688 (86.169) | 328.224 (112.684)
Statistical Analysis 1: Comparison: Participants With Obsessive-compulsive Disorder (OCD) vs Healthy Control (HC) Participants; Whole-Brain Connectome-Level Analyses were performed on the structural connectivity indices (streamline count) between 164 regions. Edge-wise structural connectivity analyses was then be conducted across the resulting matrix comprised of 164 nodes and 26,896 edges, using the Network-Based Statistics (NBS) Toolbox; Test type: Superiority — only participants were assigned to groups (OCD, HC) and we measured streamline count in these participants to index structural connectivity; p < 0.025, Regression, Linear — NBS controls for family-wise error rate using permutation testing to identify components or "clusters" of contiguous region-to-region connections. A statistical threshold of p=.025 with 10,000 permutations was used; Slope = -102.67 — Direction of comparison: HC>OCD

ADVERSE EVENTS:
Time Frame: Approximately 16-20 weeks for each participant (over 6 years and 6 months for the entire study).
Arm/Group | Participants With Obsessive-compulsive Disorder (OCD) | Healthy Control (HC) Participants
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/27
Other Adverse Events (participants affected / at risk) | 0/28 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-24): https://cdn.clinicaltrials.gov/large-docs/15/NCT02421315/Prot_SAP_000.pdf